CLINICAL TRIAL: NCT06977399
Title: The Application Value of Spectral CT in the Accurate Staging of Liver Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yunnan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KYLX2025-108
Record Dates: First submitted 2025-05-09; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The application value of spectral CT in the accurate staging of liver cancer (Experimental): Prospectively collect medical images and clinical data related to liver cancer using Philips Quark CT equipment, and evaluate the diagnostic accuracy and clinical application value in the accurate staging of liver cancer.Patients diagnosed with liver cancer in Yunnan Provincial Cancer Hospital from April 2025 to May 2026 were consecutively included, and after scanning with Philips Quark CT, the TNM stage of liver cancer patients was assessed by two radiologists, and finally statistical analysis was performed.
  Interventions: Diagnostic Test: To explore the value of spectral CT in the diagnosis and treatment of liver cancer

INTERVENTIONS:
Diagnostic Test: To explore the value of spectral CT in the diagnosis and treatment of liver cancer — The CT scan is part of the standard treatment protocol.

SUMMARY:
Spectral CT was used to prospectively collect medical images and clinical data related to liver cancer, evaluate the effect of image quality in the diagnosis of liver cancer, and evaluate the application value in the accurate staging of liver cancer, so as to provide a more accurate clinical basis for diagnosis, promote the development of individualized treatment, and ultimately improve the prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Undergo a contrast-enhanced Quark Spectral CT scan of the lower abdomen/pelvis within 1 week before treatment.
2. Age > 18 years.
3. Patients suspected of having liver cancer.
4. Patients who have signed the informed consent form.

Exclusion Criteria:

1. Severe cardiac, pulmonary, or renal insufficiency.
2. Allergy to iodine-based contrast agents.
3. Inability to cooperate with the CT examination.
4. Poor image quality of the Quark Spectral CT scan.
5. Women who are pregnant or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Pathological TNM staging | 1 day
  Pathological examination information: The pathology results using surgery/biopsy data are the gold standard, and the depth of tumor invasion, lymph node metastasis, and distant metastasis are recorded

CONTACTS AND LOCATIONS:
Overall Officials: Lianhua Ye, Study Director — Ethics Committee of Yunnan Provincial Cancer Hospital
Locations (1):
- Yunnan Cancer Hospital, Kunming, Yunnan, China